CLINICAL TRIAL: NCT02955017
Title: Use of New Technologies for the Follow-up in Adolescent Obesity
Brief Title: Mobile Health Intervention
Acronym: MHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-A00666-45
Record Dates: First submitted 2016-10-24; First posted 2016-11-04 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Obesity
Keywords: obesity; children; adolescents; new technology; mobile health; chronic disease
MeSH Terms: conditions — Obesity; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional follow-up (Active Comparator)
  Interventions: Behavioral: traditional follow_up
- Distance follow-up "new technologies" (Experimental)
  Interventions: Behavioral: distance follow-up "new technologies"

INTERVENTIONS:
Behavioral: traditional follow_up — * Multidisciplinary support with educational face to face family based intervention at 6, 9 and 12 months after inclusion.
  * Two days of a complete medical check at 9 and 15 months
  Arms: Traditional follow-up
Behavioral: distance follow-up "new technologies" — * Multidisciplinary support with long distance monitoring "Mobile apps".
  * Two days of a complete medical check at 9 and 15 months
  Arms: Distance follow-up "new technologies"

SUMMARY:
The purpose of this study is to evaluate the efficacy of a distance follow-up on body mass index decrease at 15 months compared to traditional management in obese adolescents.

DETAILED DESCRIPTION:
Childhood obesity continues to be a key challenge in France. The unit is facing a high demand with limited resources, moreover despite an intensive program of care with a multidisciplinary dedicated team, the impact on weight loss is moderate.

The hypothesis is to ameliorate results by using distance monitoring in maintenance phase.

After a traditional intensive period consisting in a weekly family-based multidisciplinary intervention, patients are randomized in two arms, traditional or distance follow-up.

Traditional follow-up is based on face-to-face multidisciplinary consultations every three months.

The distance monitoring is based on a mobile application dedicated to food behavior change and physical activity, with weekly self-monitoring, goal setting, physical activity and healthy eating support, monthly weight assessment. Pre-programmed feedbacks "motivational strategies" are included.

After one year of follow-up, adolescents are evaluated for weight loss, compliance and quality of life. The two groups will be compared.

The question is can mobile apps help to monitor and promote healthy lifestyle in obese adolescents.

ELIGIBILITY:
Inclusion Criteria:

* 11-17 years old
* Body Mass Index > 97th percentile using French reference
* Non Syndromic obesity
* Appropriate understanding of the study
* Appropriate understanding of french language, and ability in writing and reading

Exclusion Criteria:

* Mental disability, severe and uncontrolled psychiatric disorders.
* Syndromic obesity, endocrine disorders or drug-induced obesity
* Other therapeutic: bariatric surgery, medications for weight loss
* Enrolment in an other therapeutic study

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Body Mass Index Z-score | 15 months
  Body mass index z score is calculated using french reference data. success: decrease of Body Mass Index Z-score from baseline to 15 months of 0.5 standard deviation

SECONDARY OUTCOMES:
Change from baseline in mean difference of Body Mass Index Z-score between the two groups | 15 months
Percent of loss to follow-up | 15 months
Change from baseline in PedsQL score | 15 months
Change from baseline in Eating Behavior assessed by a dietitian from a questionnaire | 15 months
Change from baseline in Physical activity and sedentary behavior assessed by the number of hours of physical activity per week | 15 months
Glycemia (mmol/l) | 15 months
  Change from baseline in metabolic syndrome
Fasting insulinemia (µmol/l) | 15 months
  Change from baseline in metabolic syndrome
Homeostasis Model assessment (HOMA) | 15 months
  Change from baseline in metabolic syndrome
Dyslipidemia (mmol/l) | 15 months
  Change from baseline in metabolic syndrome
Blood pressure (mmHg) | 15 months
  Change from baseline in metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Myriam DABBAS, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Necker-Enfants malades Hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Malley G, Clarke M, Burls A, Murphy S, Murphy N, Perry IJ. A smartphone intervention for adolescent obesity: study protocol for a randomised controlled non-inferiority trial. Trials. 2014 Jan 31;15:43. doi: 10.1186/1745-6215-15-43. PMID 24485327
- [Background] Turner T, Spruijt-Metz D, Wen CK, Hingle MD. Prevention and treatment of pediatric obesity using mobile and wireless technologies: a systematic review. Pediatr Obes. 2015 Dec;10(6):403-9. doi: 10.1111/ijpo.12002. Epub 2015 Jan 12. PMID 25641770
- [Background] Svetkey LP, Batch BC, Lin PH, Intille SS, Corsino L, Tyson CC, Bosworth HB, Grambow SC, Voils C, Loria C, Gallis JA, Schwager J, Bennett GG. Cell phone intervention for you (CITY): A randomized, controlled trial of behavioral weight loss intervention for young adults using mobile technology. Obesity (Silver Spring). 2015 Nov;23(11):2133-41. doi: 10.1002/oby.21226. PMID 26530929
- [Background] Pretlow RA, Stock CM, Allison S, Roeger L. Treatment of child/adolescent obesity using the addiction model: a smartphone app pilot study. Child Obes. 2015 Jun;11(3):248-59. doi: 10.1089/chi.2014.0124. Epub 2015 Mar 11. PMID 25760813
- [Result] Foissac F, Lepage G, Briand N, Cosnefroy M, Charrat A, Dabbas M. Mobile Health Is a Cost-Effective Strategy for Managing Obesity in Adolescents: A Randomised Controlled Trial. Acta Paediatr. 2025 Dec;114(12):3233-3243. doi: 10.1111/apa.70248. Epub 2025 Jul 24. PMID 40704768